CLINICAL TRIAL: NCT02606864
Title: Non-blinded, Randomized, Single Center, Single Dose, Cross-over Study to Assess the Effect of a High Calorie/High Fat Meal on the Pharmacokinetics of Four 30 mg Nifurtimox Tablets Taken Orally by Adult Male and Female Patients Suffering From Chronic Chagas' Disease
Brief Title: Study to Assess the Food Effect on the Pharmacokinetics of Nifurtimox Tablets in Chronic Chagas' Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16005
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAYa2502 without food (Experimental): Oral intake of a single 120 mg nifurtimox dose under fasted conditions
  Interventions: Drug: Nifurtimox (BAYa2502)
- BAYa2502 with food (Experimental): Oral intake of a single 120 mg nifurtimox dose under fed conditions after ingestion of a high calorie and high fat breakfast
  Interventions: Drug: Nifurtimox (BAYa2502)

INTERVENTIONS:
Drug: Nifurtimox (BAYa2502) — Oral Intake of 4 x 30 mg nifurtimox tablets

SUMMARY:
This study will evaluate the effect of food on the absorption of the drug as well as safety and tolerability of the novel 30 mg tablet (administered as 120 mg dose) in adults suffering from chronic Chagas' disease when administered after a high-fat / high-calorie test meal (American breakfast) compared to a fasting state. This study is required as part of the clinical development of an age appropriate pediatric oral dosage form for the treatment of Chagas' disease in endemic countries according to the recommendations provided by current international guidelines (EMA Guideline on Clinical Development of Medicinal Products, EMA Note for Guidance on Oral Dosage Forms).

ELIGIBILITY:
Inclusion Criteria:

* Study participants of reproductive potential must agree to utilize two reliable and acceptable methods of contraception simultaneously when sexually active. One of these methods must include a barrier method.

Subjects who are not of reproductive potential include: vasectomized males or non-vasectomized males with documented azospermia prior to screening, as well as females who are surgically sterilized with bilateral tubal ligation or who have undergone hysterectomy. Women who are menopausal are also considered not of reproductive potential if there has been no menses > 12 months prior to screening and supported by a pre-screening follicle stimulating hormone (FSH) > 40 mIU/ml if available.

Examples of reliable and acceptable methods of birth control include, but are not limited to: diaphragm with spermicide, condoms with spermicide or oral contraception with condom use in the male partner. This applies from the signing of the informed consent up until 12 weeks after the last dose of the study medication.

* Male/female subject diagnosed with chronic Chagas' disease: Previous diagnosis of acute or chronic Chagas' disease by a health clinic prior to screening for the study. The diagnosis of chronic Chagas' disease may be made by clinical findings, supported by antibody titers if available. If there is a known history of acute disease, it is preferable to have documentation of parasites on the blood smear if available
* Age: 18 to 45 years (inclusive) at the first screening visit
* Body mass index (BMI): above/equal 18 and below/equal 29.9 kg / m²

Exclusion Criteria:

* Incompletely cured pre-existing diseases (except chronic Chagas) for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Acute Chagas'disease (During the acute phase, the parasite on a blood smear may be seen under a microscope. Different antibodies are present, depending on the course of the disease)
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Unstable or uncontrolled medical condition such as hypertension or diabetes, decompensated heart failure, gastrointestinal (GI) conditions that would interfere with the absorption of the study drug (e.g. GI ulceration, peptic ulceration, GI bleeding, gastroesophageal reflux, or other GI disease affecting gastroesophageal junction), conditions that could potentially have an impact on drug metabolism or elimination (renal, hepatic such as known hepatic or biliary abnormalities), or any clinically relevant active infections in the opinion of the investigator within 4 weeks before the screening visit, e.g. clinically relevant history or presence of significant respiratory (e.g. interstitial lung disease), hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic (e.g. diabetes), and dermatological or connective tissue disease
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them within 4 weeks before the first study drug administration, e.g. an investigational drug, any drug altering GI motility and/or gastric pH (e.g. antacids, anticholinergic, para-sympatholytics), any drug known to induce liver enzymes (e.g. dexamethasone, barbiturates, St. John's Wort [hypericum perforatum]), any drug known to inhibit liver enzymes (e.g. ketoconazole, macrolides)
* Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over 120 msec or of the QT-interval over 450 msec using Bazett's Formula (QTcB) or Fridericia's Formula (QTcF). (clinically stable subjects with Chagas'- related heart disease and pacemaker in place for >1 year and evaluated by a cardiologist ≤6 months before the first dose of study drug will not be excluded.)
* Systolic blood pressure below 100 or above 140 mmHg (after resting in supine position for a minimum of 3 min)
* Diastolic blood pressure below 50 or above 90 mmHg (after resting in supine position for a minimum of 3 min)
* Pulse rate below 45 or above 95 beats / min (after resting in supine position for a minimum of 3 min)
* Findings that would exclude the subject in the physician's judgment e.g. enlarged liver, irregular heartbeat, undiagnosed acute illness, melanoma

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the drug-concentration vs. time curve of nifurtimox from time 0 to the last data point[AUC(0-tlast)] | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24 hours
Plasma concentration nifurtimox characterized by Cmax | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24 hours
Plasma concentration of nifurtimox characterized by tmax | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24 hours
Plasma concentration of nifurtimox characterized by AUC | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24 hours

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Buenos Aires, Ciudad Auton. de Buenos Aires, Argentina